CLINICAL TRIAL: NCT03201939
Title: Optimal Management of HIV Infected Adults at Risk for Kidney Complications in Nigeria
Acronym: R3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommendations, laboratory quality control (QC) issues. All lab Q/C issues addressed; DSMB approved study re-opening, but due to length of time required to address lab QC issues, insufficient follow-up time was available to complete study.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Aminu Kano Teaching Hospital (Other); SAIC-Frederick, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, C. William Wester, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vanderbilt_University MC; U01DK112271 (NIH)
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS; Albuminuria; Kidney Diseases; Genetic Predisposition
Keywords: HIV/AIDS; sub-Saharan Africa; Kidney disease; Albuminuria; Genetic risk
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Albuminuria; Kidney Diseases; Genetic Predisposition to Disease | interventions — Lisinopril

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Medication (Intervention arm) (Active Comparator): ACE-inhibitor lisinopril
  Interventions: Drug: Lisinopril
- Placebo comparator (Control arm) (Placebo Comparator): Matched placebo
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Drug: Lisinopril — ACE-inhibitor (lisinopril)(intervention arm
  Other Names: Intervention arm
  Arms: Active Medication (Intervention arm)
Other: Placebo Oral Tablet — Comparator placebo (control arm)
  Other Names: Control arm
  Arms: Placebo comparator (Control arm)

SUMMARY:
In this study, the Investigators plan to determine the optimal means to prevent or slow the progression of kidney disease among genetically at-risk northern Nigerian HIV-infected adults. Based on data from studies of diabetic kidney disease that used medications that block the renin angiotensin aldosterone system (RAAS), we plan to evaluate whether or not RAAS inhibition (using a widely available medication that blocks RAAS) in HIV-infected adults produces similarly promising results.

DETAILED DESCRIPTION:
Individuals of African descent have a much higher risk for glomerular diseases. Specifically, there are two risk variants in the chromosome 22 APOL1 gene (G1/G2) and persons possessing 2 copies of these risk variants (G1/G1, G1/G2, or G2/G2), referred to as the high-risk (HR) genotype, are at high risk for non-diabetic kidney disease. Kopp et al. have shown that the APOL1 high-risk genotype confers sizeable odds ratios (OR) for FSGS (OR = 17), HIVAN (OR = 29 in the US; 89 in S. Africa), and hypertension-attributed end stage kidney disease (OR = 7). The presence of these risk variants is highest in West Africa, and specifically in Nigeria among persons of Hausa, Fulani, and Igbo descent. In the setting of untreated HIV infection, we have estimated that ~50% of individuals carrying the APOL1 HR genotype will develop chronic kidney disease (CKD). However, there is limited availability of dialysis and kidney transplantation in Nigeria, and most individuals will die soon after developing ESKD. Markers of kidney disease include microalbuminuria, proteinuria, and/or reduced estimated glomerular filtration rate (eGFR). All 3 have been associated with increased mortality in HIV+ adults. Increased urinary albumin excretion has diagnostic and prognostic value in the identification and confirmation of renal disease, and changes in albuminuria can be useful in assessing treatment efficacy as well as disease progression. Microalbuminuria, i.e., urine albumin to creatinine ratio (uACR) in the 30-300 mg/g range, is likely the earliest stage of CKD, analogous to diabetic microalbuminuria. The renin-angiotensin aldosterone system (RAAS) is the central player in the pathophysiology of CKD and blocking RAAS with angiotensin converting enzyme inhibitors (ACEi) is a well-recognized strategy to slow or halt renal disease progression in diabetics with CKD. To determine whether the presence of APOL1 HR genotype alters or predicts responsiveness to conventional therapy and if the addition of an ACEi to standard antiretroviral therapy (ART) reduces the risk for renal complications among West African adults, we will screen 2,600 HIV+ ART-experienced adults; to conduct the following Specific Aims:

1. To determine the prevalence of APOL1 renal risk variants and assess whether APOL1 HR status correlates with prevalent albuminuria, eGFR, and/or prevalent CKD in a West African population.
2. To assess whether RAAS inhibition (with the ACEi lisinopril) in addition to ART, compared to the existing standard-of-care (SOC), will significantly reduce the incidence of additional kidney disease manifestations. We will randomize ART-experienced (6+ months) adults with prevalent microalbuminuria (uACR 30-300 mg/g) and an eGFR of > 30 ml/min/1.73m2 to lisinopril (n=140) vs. SOC (n=140); and
3. To determine whether the APOL1 HR genotype is associated with worse longitudinal renal outcomes in Nigerians with prevalent albuminuria.

ELIGIBILITY:
Inclusion criteria:

* Participated in Study Aim 1
* 18-70 years of age
* HIV-positive (as documented by HIV-1 ELISA testing)
* On ART for a minimum of six (6) months AND having a suppressed plasma viral load result (< 20 copies/mL) within the past 6 months
* Average uACR between 30-300 mg/g (based on 2 uACRs [first morning voids], with the second obtained 4-8 weeks after the first specimen)(NOTE: All aim 1 screened patients having a uACR value > 300 mg/g will undergo urine dipstick analysis for aim 2 eligibility, and if their urine dipstick results reveals ≥ 2+ protein, then they will be considered ineligible (no additional uACR testing will be necessary to determine eligibility)
* eGFR = >60 ml/min/1.73m2 (using CKD-EPI-Cr-CyC equation) AND
* If female, non-pregnant (documentation of negative urine pregnancy test) and not breastfeeding/lactating

Exclusion criteria:

* Pregnant or currently breastfeeding
* eGFR of <60 ml/min/1.73m2 (using CKD-EPI-Cr-CyC equation)
* Average uACR > 300 mg/g (based on 2 uACRs [first morning voids], with the second obtained 4-8 weeks after the first specimen)
* K+ >5.0 meEq/L or reasons to be concerned about hyperkalemia
* Known history of Diabetes diabetes mellitus (would qualify for treatment with an ACEi/ARB)
* Poorly controlled hypertension (≥3 BP readings >160/110 in past 3 6 months)
* Known history of Congestive congestive heart failure (chronic)
* Average uACR (calculated on values obtained from 2 successive measures 4-8 weeks apart) of < 30 mg/g OR > 300 mg/g
* Relative symptomatic hypotension (BP <90/60)
* Currently receiving an ACEi and/or ARB; OR
* Lack of suitability as a study candidate (i.e. active substance use disorder, active use of potentially nephrotoxic medication(s) (i.e. traditional medicines, etc.) and/or consistent alcohol, drug, and/or traditional medication use, and/or history of poor compliance (i.e. multiple missed scheduled clinic appointments, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both males and females eligible
Enrollment: 66 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. William Wester, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Muktar H. Aliyu, MD, DrPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Investigative team will work with study biostatisticians, DSMB members, and collaborators to release analysis scripts (with publications) and devise an IPD sharing plan at/near study completion.
Time Frame: Approximately 6 months after collection of the final patient data.
Access Criteria: Deidentified data will be available after the conclusion of the study for investigators who are approved by the trial leadership at VUMC, AKTH, and NIH.

REFERENCES:
- [Background] Wudil UJ, Aliyu MH, Prigmore HL, Ingles DJ, Ahonkhai AA, Musa BM, Muhammad H, Sani MU, Nalado AM, Abdu A, Abdussalam K, Shepherd BE, Dankishiya FS, Burgner AM, Ikizler TA, Wyatt CM, Kopp JB, Kimmel PL, Winkler CA, Wester CW. Apolipoprotein-1 risk variants and associated kidney phenotypes in an adult HIV cohort in Nigeria. Kidney Int. 2021 Jul;100(1):146-154. doi: 10.1016/j.kint.2021.03.038. Epub 2021 Apr 24. PMID 33901548
- [Background] Aliyu MH, Wudil UJ, Ingles DJ, Shepherd BE, Gong W, Musa BM, Muhammad H, Sani MU, Abdu A, Nalado AM, Atanda A, Ahonkhai AA, Ikizler TA, Winkler CA, Kopp JB, Kimmel PL, Wester CW. Optimal management of HIV- positive adults at risk for kidney disease in Nigeria (Renal Risk Reduction "R3" Trial): protocol and study design. Trials. 2019 Jun 10;20(1):341. doi: 10.1186/s13063-019-3436-y. PMID 31182139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 participants were enrolled from 4/1/2021 thru 7/22/2021, with all participants being followed intensively through 11/20/2021, at which time, per DSMB recommendations, the study was paused (for reasons related to laboratory quality control (QC), specifically, the inability to accurately measure urine albumin on-site). All involved IRBs were notified and all participants were given a "Dear Participant" letter. Reasons for study pause were not at all related to any safety concerns.
Period: Overall Study
Arm/Group | Placebo Comparator (Control Arm) | Active Medication (Intervention Arm)
Started | 32 | 34
Completed | 0 | 0
Not Completed | 32 | 34
Not completed — Study was suspended by DSMB because of laboratory quality control issues. | 32 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Medication (Intervention Arm) | Placebo Comparator (Control Arm) | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (7) | 42 (6) | 42 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 32 | 66
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Nigeria | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Regression From Microalbuminuria (uACR 30-300) to Normoalbuminuria (uACR < 30 mg/g) by Study Arm
Description: Proportion of study participants regressing from microalbuminuria (uACR 30-300) to normoalbuminuria (uACR < 30 mg/g) by study arm
Time Frame: 2 years
Population: The data at 2 years was not collected since the study terminated prior to 2 years.
Arm/Group | Active Medication (Intervention Arm) | Placebo Comparator (Control Arm)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Progression From Microalbuminuria (uACR 30-300) to Macroalbuminuria (uACR > 300 mg/g) by Study Arm
Description: Proportion of study participants progressing from microalbuminuria (uACR 30-300) to macroalbuminuria (uACR > 300 mg/g) by study arm
Time Frame: 2 years
Population: The data at 2 years was not collected since the study terminated prior to 2 years.
Arm/Group | Active Medication (Intervention Arm) | Placebo Comparator (Control Arm)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Mean Change in Urinary Albumin to Creatinine Ratio (uACR)
Description: Mean change in urinary albumin to creatinine ratio (uACR) among study participants at study timepoints by study arm
Time Frame: 2 years
Population: The data at 2 years was not collected since the study terminated prior to 2 years.
Arm/Group | Active Medication (Intervention Arm) | Placebo Comparator (Control Arm)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Doubling of Serum Creatinine From Baseline
Description: Worsening renal function (as measured by serum creatinine)
Time Frame: 2 years
Population: The data at 2 years was not collected since the study terminated prior to 2 years.
Groups:
- Placebo Comparator (Control Arm): The placebo comparator includes a Matched placebo
- Active Medication (Intervention Arm): The active medication (intervention arm) includes the ACE-inhibitor lisinopril
Arm/Group | Placebo Comparator (Control Arm) | Active Medication (Intervention Arm)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: All-cause Mortality
Description: Mortality (All-cause) by study arm
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Proportion Experiencing a 40% Decline in eGFR
Description: Proportion with 40% decline in eGFR (measured using CKD-EPI-Cr-CyC equation)
Time Frame: 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Mean Change in eGFR Over Time
Description: Mean change in eGFR (measured using CKD-EPI-Cr-CyC equation)
Time Frame: 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Change in Clinical/Performance Status as Ascertained Via World Health Organization Quality of Life HIV (WHOQOL-HIV) Scale
Description: WHOQOL-HIV scale evaluates quality of life based on physical, psychological, social, environmental, and spiritual domains, as well as level of independence. We will use the 31-question version, with each question rated on a 5-point Likert scale. Scores of questions within each domain are averaged to get domain score, and final score is mean of domain scores multiplied by 4. Final score ranges from 4 to 20, with 20 being optimal.
Time Frame: Baseline, 1 year, 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Change in Clinical/Performance Status as Ascertained Via Karnofsky Performance Score
Description: Karnofsky Performance Score measures change in clinical/performance status with values ranging from 0 to 100, where 100 is perfect health and 0 is death.
Time Frame: Baseline, 1 year, 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE data was collected over 7 months; NOTE: AE data planned to be collected among all study participants for the full 2 years of study follow-up, but study was suspended early due to identified laboratory quality issues (per DSMB) and once these lab QA/QC issues were rectified, there was insufficient time to follow all study participants for full, specified duration of follow-up; therefore the study was terminated.
Groups:
- Placebo Comparator (Control Arm): Placebo comparator (Control arm) -- matched placebo
- Active Medication (Intervention Arm): Active study medication -- ACE-inhibitor lisinopril
Arm/Group | Placebo Comparator (Control Arm) | Active Medication (Intervention Arm)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 3/32 | 5/34
Other Adverse Events (participants affected / at risk) | 11/32 | 21/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Comparator (Control Arm) (N=32) | Active Medication (Intervention Arm) (N=34)
Angioedema (Vascular disorders) | 0 | 1
Worsening Kidney Function, decrease in eGFR and/or uACR (Renal and urinary disorders) | 3 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Comparator (Control Arm) (N=32) | Active Medication (Intervention Arm) (N=34)
Hypotension (Cardiac disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dizziness (General disorders) | 0 | 2
Hyperkalemia (Investigations) | 0 | 1
Headache (General disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hypertension (Cardiac disorders) | 4 | 2
Fever (General disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Emesis (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Upper/Lower Limb Pain (General disorders) | 0 | 2
Hypokalemia (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
The primary limitation of this study was laboratory quality control (QC) issues. While all QC concerns were addressed, the time required to resolve them led to a delay in the study. Although the Data and Safety Monitoring Board (DSMB) approved the study's re-opening, the extended resolution period resulted in insufficient follow-up time to complete the study as originally planned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03201939/Prot_SAP_000.pdf